CLINICAL TRIAL: NCT00423150
Title: A Phase 2 Study of Temozolomide (SCH 52365) in Subjects With Advanced Aerodigestive Tract Cancers Selected for Methylation of O6-Methyl-Guanine-DNA Methyltransferase (MGMT) Promoter
Brief Title: Phase 2 Study of Temozolomide in Pre-Selected Advanced Aerodigestive Tract Cancers (Study P04273AM2)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04273
Record Dates: First submitted 2006-11-30; First posted 2007-01-18 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Neoplasm; Head and Neck Neoplasm; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide capsules 150 mg/m^2 daily on a 7-day on / 7-day off schedule for each 28-day cycle, until disease progression, intolerable toxicity, or withdrawal of consent.
  Other Names: Temodal, TMZ, SCH 52365

SUMMARY:
This study is proposed to evaluate the efficacy and safety of temozolomide, an oral anti-cancer agent, in a participant population selected for a biomarker. Participants with colorectal cancer, non-small-cell lung cancer, head and neck cancer, or esophageal cancer will be included.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age.
* Participants must have metastatic colorectal cancer (CRC), recurrent or metastatic head & neck (H&N) or esophageal cancer, or locally advanced, inoperable, or metastatic non-small cell lung cancer (NSCLC).
* Participants must have a tumor sample or a blood sample tested positive for the presence of the biomarker.
* Participants may have up to 3 prior regimens for CRC, up to 3 prior regimens for NSCLC, up to 2 prior regimens for H&N and esophageal cancer.
* Participants must have at least one measurable lesion.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Participants must have adequate hematologic, renal, and liver functions.
* Participants must be able to take the study medication capsules orally, or through a feeding tube without the capsules being opened.
* Participants of childbearing potential must agree to use a medically accepted method of contraception.

Exclusion Criteria:

* Participants who have received treatment for a second malignancy within 1 year before screening, and are considered to be at risk of relapse within 1 year after screening.
* Participants with unstable or progressing central nervous system (CNS) metastasis. Participants with known CNS metastasis may be included if a) the subject is asymptomatic, b) there is no requirement for steroids or antiseizure medications, or the required doses are stable, and c) there is no associated midline shift or (in the opinion of the investigator) significant edema.
* Participants who received prior temozolomide or dacarbazine treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-01-26 (Actual); Primary Completion 2009-06-11 (Actual); Study Completion 2009-06-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hochhauser D, Glynne-Jones R, Potter V, Gravalos C, Doyle TJ, Pathiraja K, Zhang Q, Zhang L, Sausville EA. A phase II study of temozolomide in patients with advanced aerodigestive tract and colorectal cancers and methylation of the O6-methylguanine-DNA methyltransferase promoter. Mol Cancer Ther. 2013 May;12(5):809-18. doi: 10.1158/1535-7163.MCT-12-0710. Epub 2013 Feb 26. PMID 23443801

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide: Temozolomide capsules 150 mg/m^2 daily on a 7-day on/7-day off schedule for each 28-day cycle. Temozolomide is the only treatment group, and and all participants received the same dosing regimen.
Period: Overall Study
Arm/Group | Temozolomide
Started | 86
Completed | 0
Not Completed | 86
Not completed — Adverse Event | 11
Not completed — Progression of disease being studied | 69
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance with protocol | 1
Not completed — Administrative | 4

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Tumor Responses (Complete and Partial Response)
Description: Tumor response rate was based on Response Evaluation Criteria in Solid Tumors (RECIST).
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: From start of treatment until participant's disease progression, intolerable toxicity or death, which ever comes first
Population: Population for the primary outcome measure is all evaluable participants per protocol definition (82 participants).
  Complete response is defined as disappearance of all target lesions.
  Partial response is defined as at least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Measure: Number; unit: Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 82
Participants
  Number of participants with Complete Response | 0
  Number of participants with Partial Response | 5

ADVERSE EVENTS:
Description: Other adverse events: these non-serious events are treatment-emergent.
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 37/86
Other Adverse Events (participants affected / at risk) | 83/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=86)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (7)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (4)
FATIGUE (General disorders) | 2 (2)
MULTI-ORGAN FAILURE (General disorders) | 1 (1)
PYREXIA (General disorders) | 3 (3)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (2)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
BLOOD UREA INCREASED (Investigations) | 1 (2)
OXYGEN CONSUMPTION INCREASED (Investigations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
CEREBRAL ARTERY THROMBOSIS (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (6)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NEPHROSTOMY TUBE REMOVAL (Surgical and medical procedures) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=86)
ANAEMIA (Blood and lymphatic system disorders) | 17 (30)
LYMPHOPENIA (Blood and lymphatic system disorders) | 9 (18)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 19 (55)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (13)
CONSTIPATION (Gastrointestinal disorders) | 22 (25)
DIARRHOEA (Gastrointestinal disorders) | 21 (37)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (8)
NAUSEA (Gastrointestinal disorders) | 45 (84)
VOMITING (Gastrointestinal disorders) | 35 (53)
ASTHENIA (General disorders) | 10 (13)
FATIGUE (General disorders) | 36 (75)
OEDEMA PERIPHERAL (General disorders) | 7 (10)
PYREXIA (General disorders) | 7 (13)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6)
PLATELET COUNT DECREASED (Investigations) | 5 (9)
WEIGHT DECREASED (Investigations) | 13 (13)
ANOREXIA (Metabolism and nutrition disorders) | 31 (33)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 7 (11)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5 (9)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (6)
DIZZINESS (Nervous system disorders) | 11 (16)
HEADACHE (Nervous system disorders) | 13 (27)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 6 (6)
ANXIETY (Psychiatric disorders) | 5 (5)
INSOMNIA (Psychiatric disorders) | 7 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (12)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 (9)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (8)
RASH (Skin and subcutaneous tissue disorders) | 12 (17)
HYPOTENSION (Vascular disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
Due to low response rate for colorectal cancer in interim analyses, low enrollment in head & neck and non-small cell lung cancer groups due to low methylation rates, and low overall response rate in esophageal cancer group, the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results

of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor, 45 days prior to submission, review copies of abstracts or manuscripts for publication that report any results of the study. If the parties disagree, investigator agrees to meet with the sponsor, prior to submission, for the purpose of making good faith efforts to discuss/resolve any such issues.